CLINICAL TRIAL: NCT01166971
Title: A Randomized, Subject-masked Comparison of Visual Function After Bilateral Implantation of Presbyopia-correcting IOLs
Brief Title: A Comparison of Visual Function After Bilateral Implantation of Presbyopia-correcting Intraocular Lenses (IOLs)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: M09-050
Record Dates: First submitted 2010-07-19; First posted 2010-07-21 (Estimated); Results first posted 2011-11-08 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2011-11

CONDITIONS: Cataract
Keywords: presbyopia; intraocular lens
MeSH Terms: conditions — Cataract; Presbyopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ReSTOR +3 (Experimental): Bilateral Implantation of ReSTOR +3 Intraocular lenses after cataract extraction
  Interventions: Device: ReSTOR +3
- Tecnis MF (Active Comparator): Bilateral Implantation of Tecnis Multifocal Intraocular lenses after cataract extraction
  Interventions: Device: Tecnis MF

INTERVENTIONS:
Device: ReSTOR +3 — Bilateral implantation of ReSTOR +3 Intraocular Lenses (IOLs) after cataract extraction
  Arms: ReSTOR +3
Device: Tecnis MF — Bilateral implantation of Tecnis Multifocal (MF) Intraocular Lenses (IOLs) after cataract extraction
  Arms: Tecnis MF

SUMMARY:
The purpose of this study is to prospectively evaluate postoperative visual and refractive parameters in a series of subjects bilaterally implanted with the AcrySof® IQ ReSTOR® +3 versus those bilaterally implanted with the Tecnis Multifocal 1-piece.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with bilateral cataracts
* candidate for presbyopic lens

Exclusion Criteria:

* >1 Diopter (D) preoperative astigmatism by Keratometry (K)readings
* pre-existing conditions that could skew the results

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2010-07; Primary Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - The Eye Center of North Florida, Panama City, Florida
  - Carolina Eye Care Physicians, Charleston, South Carolina
  - Whitsett Vision Group, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Bilateral diagnosis of cataracts of subjects >21 years of age
Pre-assignment Details: During the preoperative exam, subjects were examined to ensure they met the inclusion/exclusion criteria.
Period: Overall Study
Arm/Group | ReSTOR +3 | Tecnis MF
Started | 33 | 31
Completed | 32 | 30
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ReSTOR +3 | Tecnis MF | Total
Number analyzed (Participants) | 33 | 31 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 10 | 29
  >=65 years | 14 | 21 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 38
  Male | 15 | 11 | 26

OUTCOME MEASURES:

1. Primary Outcome: Defocus Curve
Description: A defocus curve is created by multiple measurements of one's visual acuity at different spherical powers (recorded as Diopters (D)). Visual Acuity (VA) is measured in logMAR. LogMAR is the "logarithm of the minimum angle of resolution".
Time Frame: 3 months after surgery
Population: In the ReSTOR +3 population, 1 subject did not complete the assessment at -5.00 D; therefore, only 32 subjects were used for this measure.
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | ReSTOR +3 | Tecnis MF
Number analyzed (Participants) | 33 | 29
LogMAR
  -5.00 Diopter (D) | 0.585 (0.204) | 0.653 (0.116)
  -4.50 D | 0.490 (0.204) | 0.475 (0.115)
  -4.00 D | 0.388 (0.189) | 0.337 (0.107)
  -3.50 D | 0.261 (0.183) | 0.168 (0.114)
  -3.00 D | 0.126 (0.185) | 0.046 (0.104)
  -2.50 D | 0.017 (0.144) | 0.073 (0.113)
  -2.00 D | 0.055 (0.147) | 0.222 (0.178)
  -1.50 D | 0.245 (0.175) | 0.326 (0.120)
  -1.00 D | 0.212 (0.144) | 0.225 (0.128)
  -0.50 D | 0.052 (0.132) | 0.072 (0.120)
  0.00 D | -0.048 (0.097) | -0.044 (0.085)
  0.50 D | 0.035 (0.112) | 0.032 (0.111)
  1.00 D | 0.258 (0.140) | 0.237 (0.200)
  1.50 D | 0.434 (0.153) | 0.364 (0.176)
  2.00 D | 0.539 (0.168) | 0.446 (0.136)

ADVERSE EVENTS:
Time Frame: Adverse events were collected at all study visits.
Arm/Group | ReSTOR +3 | Tecnis MF
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/30
Other Adverse Events (participants affected / at risk) | 0/32 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The existence of this clinical study is confidential and should not be discussed with persons outside of the study. You shall hold confidential, and not disclose directly or indirectly to any third party other than those persons involved in the study who have a need to know, the protocol, the data arising out of the study, and any other information related to the study or to Alcon's products or research programs that is provided by Alcon to you (the "Confidential Information").